CLINICAL TRIAL: NCT00400309
Title: A Double Blind, Controlled, Randomised, Clinical Study to Assess the Safety of Repevax® Administered One Month After Revaxis® or Placebo to Healthy Adults
Brief Title: Safety of REPEVAX® Given One Month After REVAXIS®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: F06-Td5I-301
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Healthy Adult

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- REPEVAX® after REVAXIS® (Experimental): REVAXIS® at Visit 1 (Day 0) and REPEVAX®) at Visit 2 (Day 28).
  Interventions: Biological: REPEVAX® after REVAXIS®
- REPEVAX® after Placebo (Active Comparator): Placebo at Visit 1 (Day 0) and REPEVAX®) at Visit 2 (Day 28).
  Interventions: Biological: REPEVAX® after Placebo

INTERVENTIONS:
Biological: REPEVAX® after REVAXIS® — Tetanus, diphtheria, tetanus, pertussis (acellular, component) and poliomyelitis (inactivated) vaccine after tetanus, diphtheria, poliomyelitis (inactivated)
  Arms: REPEVAX® after REVAXIS®
Biological: REPEVAX® after Placebo — Tetanus, diphtheria, tetanus, pertussis (acellular, component) and poliomyelitis (inactivated) vaccine after placebo
  Arms: REPEVAX® after Placebo

SUMMARY:
Primary objective:

* To describe the safety profile of a Tetanus, Diphtheria, Poliomyelitis and Pertussis vaccine (REPEVAX®) when administered as a pertussis booster 1 month after a Tetanus, Diphtheria, Poliomyelitis vaccine (REVAXIS®) as compared to the safety profile of REPEVAX® administered one month after Placebo.

Secondary objectives:

* To describe the safety of Td-IPV vaccine (REVAXIS®) or Placebo administered to healthy adults.
* To describe the safety of TdaP-IPV vaccine (REPEVAX®) administered one month after Td-IPV vaccine (REVAXIS®) or one month after Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult, with vaccination history (by written evidence) of a minimum of 5 doses of a tetanus, diphtheria and poliomyelitis containing vaccine as recommended in the French vaccination calendar at 18 years old, and a maximum of 8 doses.
* Last dose of a tetanus and/or diphtheria and/or poliomyelitis containing vaccine administered either alone or in combination at least 5 years prior to the administration of the first study vaccine.

Exclusion Criteria:

* Prior known hypersensitivity reaction to any diphtheria and/or tetanus and/or poliomyelitis and/or pertussis containing vaccine
* Any current (≤ 3 days) significant underlying disease or acute febrile illness (oral temperature ≥37.5°C)
* Known immunological deficiency
* Known malignant disease
* Known neurological disorder
* Any long-term (≥ 14 days) non steroid anti-inflammatory therapy given daily within the previous 30 days
* Known history of severe thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection
* Any previous (≤ 90 days) administration of blood-derived products or immunoglobulins or scheduled to be administered through Visit 3
* Any recent administration (≤ 30 days) of a vaccine or scheduled vaccination

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
injection sites reactions and systemic events during the 7 day-safety period post-vaccination with TdaP-IPV vaccine. | 7 days

SECONDARY OUTCOMES:
injection-site adverse reactions and systemic adverse events during the 14 day-safety period post-vaccination with Td-IPV vaccine, TdaP-IPV vaccine and placebo and serious adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (4):
- France (4):
  - Clermont-Ferrand
  - Lyon
  - Montpellier
  - Paris